CLINICAL TRIAL: NCT02160054
Title: Specified Drug Use-Results Survey of Graceptor® Capsules 0.5mg, 1 mg, and 5 mg in Kidney Transplant Patients
Brief Title: Specified Drug Use-results Survey of Graceptor in Patients With Kidney Transplantation (Switching From Cyclosporine)
Status: Completed | Type: Observational
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: GRA006
Record Dates: First submitted 2014-06-09; First posted 2014-06-10 (Estimated); Last update posted 2024-10-21 (Actual); Status verified 2019-04

CONDITIONS: the Maintenance Phase After Kidney Transplantation
Keywords: tacrolimus; cyclosporine; Graceptor®; kidney transplantation
MeSH Terms: interventions — Tacrolimus

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1: patients with kidney transplantation who converted the immunosuppressant from cyclosporine to Graceptor ®
  Interventions: Drug: Graceptor®

INTERVENTIONS:
Drug: Graceptor® — oral
  Other Names: tacrolimus; FK506

SUMMARY:
To evaluate the safety and efficacy of Graceptor ® in patients with kidney transplantation when converted from cyclosporine

ELIGIBILITY:
Inclusion Criteria:

* Patients who are converted to Graceptor® from cyclosporine in the maintenance phase after kidney transplantation.
* Patients who meet one or more of following criteria

  1. Decrease in kidney function: GFR (or eGFR) less than 60 mL/min, or investigator's decision
  2. Hypertension: systolic/diastolic blood pressure 130/80 mmHg or more or treatment with an antihypertensive drug
  3. Hyperlipidaemia: LDL cholesterol 120 mg/dL or more, or treatment with an antihyperlipidemic drug
  4. Rejection: antibody mediated rejection by Banff classification borderline changes or more severe, or investigator's decision
  5. Other adverse events and patients who cannot continue cyclosporine treatment based on investigator's decision

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who are converted to Graceptor® from cyclosporine in the maintenance phase after kidney transplantation.
Sampling Method: Non-Probability Sample
Enrollment: 289 (Actual)
Dates: Start 2013-11-15 (Actual); Primary Completion 2016-03-31 (Actual); Study Completion 2016-03-31 (Actual)

PRIMARY OUTCOMES:
Rate of treatment continuation (incidence of rejection, death, graft loss, or adverse event) | 12 months

SECONDARY OUTCOMES:
Renal function, hypertension, hyperlipidaemia, other adverse events | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Use Central Contact, Study Director — Astellas Pharma Inc
Locations (30):
- Japan (30):
  - Site JP00010, Numakunai, Iwate
  - Site JP00001, Aichi
  - Site JP00015, Chiba
  - Site JP00003, Ehime
  - Site JP00029, Fukuoka
  - Site JP00009, Fukushima
  - Site JP00017, Gifu
  - Site JP00002, Hiroshima
  - Site JP00005, Hokkaido
  - Site JP00024, Hyōgo
  - Site JP00012, Ibaraki
  - Site JP00020, Ishikawa
  - Site JP00026, Kagawa
  - Site JP00030, Kagoshima
  - Site JP00014, Kanagawa
  - Site JP00027, Kochi
  - Site JP00028, Kumamoto
  - Site JP00008, Kyoto
  - Site JP00019, Mie
  - Site JP00011, Miyagi
  - Site JP00006, Nagasaki
  - Site JP00023, Nara
  - Site JP00013, Niigata
  - Site JP00025, Okayama
  - Site JP00022, Osaka
  - Site JP00016, Saitama
  - Site JP00018, Shizuoka
  - Site JP00007, Tokyo
  - Site JP00021, Wakayama
  - Site JP00004, Yamagata

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.